CLINICAL TRIAL: NCT06323421
Title: Mindfulness and CRC Risk Factor Reduction: Targeting Chronic Stress For Colorectal Cancer Risk Factor Reduction A Pilot Feasibility Study Among Vulnerable At-Risk Black Females
Brief Title: Targeting Chronic Stress for Reducing Risk Factors for Colorectal Cancer
Acronym: MindCRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Lisa Tussing-Humphreys, Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY2023-1359
Record Dates: First submitted 2024-03-01; First posted 2024-03-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Mindfulness; Colon Cancer; Females
MeSH Terms: conditions — Colonic Neoplasms | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Experimental): 8-week group and individual mindfulness training and practice
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Participants attend seven 60-90 min group mindfulness sessions each week and a 1/2 day retreat, with three sessions in-person and six sessions remote, led by a mindfulness interventionist. Additionally, participants will be encouraged to engage for at least 30 minutes per week in asynchronous mindfulness activities through a web-based program to increase exposure to mindfulness practices beyond group sessions.

SUMMARY:
Many neighborhoods in Chicago experience daily exposure to stressors including economic inopportunity and violent crime in public spaces. There is mounting evidence that chronic psychosocial stress can facilitate carcinogenesis by modulating the gut microbiome and immune system. The proposed research aims to study the practice of mindfulness to mitigate CPS and reduce colorectal cancer risk factors among Black American women at elevated risk.

DETAILED DESCRIPTION:
Chronic stress can directly and indirectly promote carcinogenesis through immune, metabolic, and microbial pathways. Our overarching hypothesis is that reducing chronic stress will have important implications for colon cancer risk reduction among vulnerable and high-risk populations. A promising approach for reducing chronic stress is mindfulness practices. Mindfulness is a meditation-based technique to achieve a state of mind used to experience higher awareness or consciousness. We propose to pilot test an 8-week Mindfulness intervention delivered in a hybrid format (synchronous and asynchronous sessions) among 40 Black females at elevated risk of colon cancer, who reside in vulnerable communities and who report moderate to high perceived stress. At baseline and post-intervention, participants will provide blood and stool undergo body composition analysis, and complete mood and lifestyle-related surveys. The specific aims are to: test the feasibility and acceptability of the intervention and evaluate the preliminary effect on stress and weight, fasting glucose, inflammation markers, and the gut microbiome - risk markers and risk pathways associated with colon tumorigenesis. While relieving social stressors is the paramount goal, addressing chronic stress at the individual level is achievable now, with implications for CRC risk reduction. If successful, data generated here will serve in developing a fully powered trial to test if MBSR is efficacious for CRC risk reduction among high-risk vulnerable populations in Chicago.

ELIGIBILITY:
Inclusion Criteria:

* Female based on sex assigned at birth
* Self-identify as Black
* Age 45-65 years old
* Completed a colonoscopy in the past 24 months,
* Classify as elevated risk of CRC defined as: any colorectal adenoma detected in past 24 months
* Own and use a smartphone, computer, or tablet with access to the Internet
* Score ≥ 14 on the PSS at screening
* Reside in a Chicago community with high violent crime

Exclusion Criteria:

* History of CRC
* Antibiotics (oral/IV) in the past 2 months
* Inflammatory bowel disease or genetic predisposition to CRC
* Cancer diagnosis or cancer treatment in the past 12 months
* Consume > 50 grams of ethanol daily
* Use combustible tobacco
* Bariatric surgery or bowel resection
* Immunodeficiency/autoimmune disease
* Uncontrolled diabetes (HbA1c > 9% based on EHR)
* Fiber or pre-/probiotic supplements > 3 days per week
* Serrated adenoma at the recent colonoscopy given the molecular features are distinct
* Significant health conditions or take medications that impact participation or expected outcomes (e.g., β-blocker, Cushing's syndrome, and corticosteroids - inhaled, topical, oral in the past month given effects on hair cortisol measurement)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility measures | Monitored across the duration of study and 8-week intervention
  easible if ≥ 30% of those approached enroll at a minimum rate of 1-3 women/week for each wave and ≥ 80% of women enrolled are retained with complete data collection at both assessment time-point
Acceptability | Week 4 and post-intervention at week 9
  The intervention will be deemed acceptable if women attend ≥ 80% of the Mindfulness group sessions, engage with ≥ 80% of the asynchronous Mindfulness content and score ≥ 16 on the acceptability survey.

OTHER OUTCOMES:
Body mass index | Baseline and post-intervention at week 9
  weight in kg divided by height in meters squared
Stress measure | Baseline and post-intervention at week 9
  Hair cortisol concentration
Fasting glucose | Baseline and post-intervention at week 9
  Measured in serum
Gut microbiota composition | Baseline and post-intervention at week 9
  16S rRNA amplicon sequencing from stool
Gut inflammation | Baseline and post-intervention at week 9
  Fecal calprotectin
Adiposity | Baseline and post-intervention at week 9
  % body fat and visceral body fat area from whole body DEXA
Epinephrine | Baseline and post-intervention at week 9
  From serum measured via mass spectrometry
Norepinephrine | Baseline and post-intervention at week 9
  From serum measured via mass spectrometry
Cortisol | Baseline and post-intervention at week 9
  From serum measured via mass spectrometry
Resting heart rate | Baseline and post-intervention at week 9
  Measured with an electronic monitor
Blood lipids | Baseline and post-intervention at week 9
  From serum - total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides
Fasting insulin | Baseline and post-intervention at week 9
  From serum
Hemoglobin A1c | Baseline and post-intervention at week 9
  From whole blood
Systemic inflammation | Baseline and post-intervention at week 9
  C-reactive protein measured in serum

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No